CLINICAL TRIAL: NCT06383559
Title: Safety and Efficacy of XELOX Combined With Sintilimab and Lenvatinib in Advanced AFP-positive Gastric Cancer Patients, a Multi-center, Prospective, Single-arm Phase II Trial
Brief Title: Safety and Efficacy of XELOX Combined With Sintilimab and Lenvatinib in Advanced AFP-positive Gastric Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJMUCH-GI-GC07
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — lenvatinib; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): XELOX regimen combined with Sintilimab and Lenvatinib
  Interventions: Drug: Lenvatinib and Sintilimab

INTERVENTIONS:
Drug: Lenvatinib and Sintilimab — XELOX regimen combined with Sintilimab and Lenvatinib

SUMMARY:
This is a multi-center, prospective, open label phase 2 study evaluating the safety and efficacy of standard first-line chemotherapy XELOX regimen combined with Sintilimab (anti-PD-1 antibody) and Lenvatinib in the treatment of advanced AFP-positive gastric cancer. This study was conducted in the Department of Gastrointestinal Medical Oncology, Tianjin Medical University Cancer Institute and Hospital. Previous phase 1 dose escalation study (TJMUCH-GI-GC002) has demonstrated that such combinational pattern was well tolerated with promising efficacy. In this study, patients with AFP-positive and HER-2-negative advanced gastric cancer who had not received palliative systematic treatment in the past will be enrolled. Patients who met the inclusion criteria were treated with XELOX regimen combined with Sintilimab plus Lenvatinib every 3 weeks until disease progression or intolerable adverse reactions or death. The treatment regimen is XELOX chemotherapy (oxaliplatin 130mg/ m2, d1, capecitabine 850-1250 mg/m2, bid, d1-14, every 3 weeks) in combination with Sintilimab (>=60kg, 200 mg; <60kg, 3mg/kg; intravenous infusion, every 3 weeks) plus Lenvatinib (determined from previous phase 1 study, 16mg, orally once a day). Patients received regular and periodic reviews, with imaging evaluations every 6 weeks. Safety will be evaluated by AE and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years old;
2. Patients with advanced / metastatic gastric cancer diagnosed by histopathology, without liver like differentiation, HER-2 negative, AFP ≥ 20ng / ml;
3. No previous palliative systemic treatment;
4. There are measurable metastatic lesions according to RECIST version 1.1;
5. ECOG physical status score is 0 or 1；
6. Normal organ function: Neutrophil count ≥ 1.2 × 109/L, Platelet count ≥ 100 × 109/L, Hemoglobin (HB) ≥ 80g/L, Total bilirubin ≤ 1.5mg/dl, AST and ALT ≤ 100 IU/L. If the abnormal liver function is due to liver metastasis, AST and ALT should be ≤ 200 IU/L, Creatinine ≤ 1.5 times* upper limit of normal, International standardization ratio (INR) ≤ 1.5;
7. Urinary protein: meet one of the following conditions Urinary protein (test paper method) is 2 + or less, Urinary protein/creatinine (UPC) ratio < 3.5, Determination of 24-hour urinary protein, urinary protein ≤ 3500mg;
8. Before receiving treatment, the patient has recovered the adverse events related to chemotherapy, radiotherapy and surgery to grade 1 or below (CTCAE 5.0);
9. For women with fertility potential with negative pregnancy test within 14 days before enrollment, male and female patients should agree to use appropriate contraceptive methods from the beginning of the first treatment to 120 days after the last treatment;
10. Patients who can take oral drugs;
11. Signed the informed consent.

Exclusion Criteria:

* 1. Patients who received surgery and radiotherapy within 2 weeks before enrollment; 2. Patients who have previously been treated with Lenvatinib or any anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs; 3. Patients with uncontrollable hypertension (systolic blood pressure ≥ 160mmHg and diastolic blood pressure ≥ 90mmHg); 4. Patients with acute coronary syndrome (including myocardial infarction and unstable angina) who had undergone coronary angioplasty within 6 months before enrollment; 5. Patients with symptomatic brain metastases; 6. Patients with New York Heart Association (NYHA) grade II or above congestive heart failure or severe arrhythmia with severe cardiovascular damage in the past 6 months; 7. The patients had active malignancies in the past 24 months (except for melanoma in situ, basal cell carcinoma of the skin or squamous cell carcinoma or carcinoma in situ of the cervix) 8. The patients have severe (hospitalized) complications 9. Patients with a history of gastrointestinal perforation and/or gastrointestinal fistula within 6 months before enrollment; 10. Patients with active hepatitis; 11. Patients with a history of human immunodeficiency virus (HIV) infection; 12. Patients with symptoms or signs of active interstitial pulmonary disease; 13. Patients with autoimmune diseases or a history of chronic or recurrent autoimmune diseases; 14. Patients who need systemic corticosteroids (excluding temporary use for testing, prophylactic administration of allergic reactions or reduction of swelling associated with radiotherapy) or immunosuppressants, or patients who receive such treatment within 14 days before enrollment; 15. The patient has a history of (non-infectious) pneumonia requiring steroids or has a current history of pneumonia; 16. Patients who received live vaccine < 30 days before starting trial drug treatment; The patient has serious non-healing wounds, ulcers or fractures; 17. Pregnant or lactating women; 18. The investigator determined that the patient is not suitable to be the subject of this trial; 19. Other circumstances that the investigator considers inappropriate to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  the rate of patients with PR and CR

SECONDARY OUTCOMES:
OS | 24 months
  The time from the beginning of treatment to the time when the patient dies from any cause
PFS | 24 months
  The time from the beginning of treatment to the time when the disease progresses or the patient dies from any cause

OTHER OUTCOMES:
AE | 24 months
  Safety will be evaluated by AE

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No